CLINICAL TRIAL: NCT06480162
Title: Impact of Mechanical Ventilation on Hippocampal Oscillation and Respiratory-hippocampus Coupling
Brief Title: Mechanical Ventilation on Hippocampus
Status: Recruiting | Type: Observational
Sponsor: Beijing Sanbo Brain Hospital (Other)
Responsible Party: Principal Investigator, Zhonghua Shi, MD, PhD, Deputy president of the department ICU, Beijing Sanbo Brain Hospital
Other Study IDs: VABI-Hipp
Record Dates: First submitted 2024-04-27; First posted 2024-06-28 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-06

CONDITIONS: Mechanical Ventilation Complication; Brain Injuries
Keywords: Ventilator Associated Brain Injury; Hippocampus Oscillation; Mechanical Ventilation
MeSH Terms: conditions — Brain Injuries | interventions — Respiration, Artificial

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Mechanical ventilation — After replacing the electrode, we'll monitor the EEG activity of the hippocampus and other cortex regions while weaning off mechanical ventilation.

SUMMARY:
Ventilator-associated brain injury (VABI) frequently occurs in ICU patients. Although animal studies indicate the hippocampus as a key target of VABI, its relevance in human patients remains uncertain. In this study, the investigators aim to monitor hippocampal EEG activity during the weaning process of patients off mechanical ventilation, and also exploring the coupling between breathing patterns and hippocampal activity.

DETAILED DESCRIPTION:
[Rational] Although mechanical ventilation (MV) is crucial for saving lives, the high incidence of ventilator-associated brain injury (VABI) in ICU patients, affecting up to 80% of cases, raises significant clinical concerns. VABI not only increases mortality and morbidity rates but also strains healthcare resources. Despite abundant evidence from preclinical studies, the precise impact of mechanical ventilation on humans remains largely unknown. Understanding these effects is crucial for uncovering the mechanisms behind VABI and subsequently preventing and treating this complication.

[Methods] Patients with drug-resistant epilepsy scheduled for stereoelectroencephalography (sEEG) exploration as part of their pre-surgical assessment will undergo eligibility screening. During the study, sEEG signals and respiratory data will be simultaneously collected from the hippocampus and other relevant limbic structures under various mechanical ventilation scenarios. These scenarios include controlled ventilation at different levels of positive end-expiratory pressure (PEEP, 5cmH2O vs. 10cmH2O) and respiratory rates (RR, 10 vs. 20 bpm), assisted ventilation, and natural breathing phases. Following the discontinuation of mechanical ventilation, patients will be monitored for up to 7 days to evaluate the occurrence of delirium. Additionally, simultaneous intracranial EEG recordings from relevant cortical and subcortical regions will be conducted.

[Aims] The current study aims to investigate the effects of mechanical ventilation, including variations in RR and PEEP, on neurophysiological electrical oscillations within the hippocampus, as well as the relationship between breathing patterns and hippocampal activity. Furthermore, the investigators will explore the impact of mechanical ventilation on other cortical areas involved in breathing, depending on electrode positioning, and examine the interactions between these brain regions and the hippocampus.

ELIGIBILITY:
Inclusion Criteria:

* Age: ≥ 18 years
* ASA: I - II
* w/ electrode inside hippocampus (≥ 1 contacts)
* Singed consent form

Exclusion Criteria:

* Seizure occurrence ≤ 36 hours before op.
* Structural brain damage
* History of using: opioids, enzyme-inducing medications, sleep aids, or excessive alcohol consumption
* History of mechanical ventilation (>24h)
* Cognitive impairment
* Operation within 6 months
* Participate in other clinical trials in the last four weeks
* Pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with drug-resistant epilepsy and scheduled for sterero-electroencephalograophy (sEEG) exploration as part of pre-surgical assessment will be screened for eligibility.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2024-05-08 (Actual); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
intracranial EEG (iEEG) recording of the hippocampus | During the process of weaning off mechanical ventilation, assessed up to 3 hours.
  The iEEG data from each patient will be analyzed using Python (version 3.12.4). The data will be represented as power spectral density, also known as the power spectrum or spectrum, which measures the frequency distribution of energy or power within a signal. The power spectrum for each channel will be computed using the Fast Fourier Transform (FFT).

CONTACTS AND LOCATIONS:
Overall Officials: Zhonghua Shi, PhD,MD, Principal Investigator — Capital Medical University
Locations (1):
- Beijing Sanbo Brain Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No